CLINICAL TRIAL: NCT04854668
Title: A Randomized, Open-label, Parallel Controlled, Multi-center Phase III Study of Anlotinib Hydrochloride Capsule Combined With Chemotherapy as First-line Treatment in Subjects With RAS/BRAF Wild Metastatic Colorectal Cancer
Brief Title: A Study of Anlotinib Hydrochloride Capsule Combined With Chemotherapy as First-line Treatment in Subjects With RAS/BRAF Wild Metastatic Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALTN-Ⅲ-02
Record Dates: First submitted 2021-04-21; First posted 2021-04-22 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anlotinib + CapeOx (Experimental): Anlotinib combined with CapeOx(Oxaliplatin+Capecitabine) were used for 4-8 cycles, each cycle is 3 weeks. After 8 cycles, the regimen is changed to Anlotinib combined with Capecitabine.
  Interventions: Drug: Anlotinib hydrochloride capsule; Drug: Oxaliplatin; Drug: Capecitabine
- Bevacizumab + CapeOx (Active Comparator): Bevacizumab combined with CapeOx(Oxaliplatin+Capecitabine) were used for 4-8 cycles, each cycle is 3 weeks. After 8 cycles, the regimen is changed to Bevacizumab combined with Capecitabine.
  Interventions: Drug: Bevacizumab; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Anlotinib hydrochloride capsule — Anlotinib hydrochloride capsule 12mg given orally in fasting conditions, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21)；
  Arms: Anlotinib + CapeOx
Drug: Bevacizumab — Bevacizumab 7.5mg/kg, intravenous drip, on Day 1
  Arms: Bevacizumab + CapeOx
Drug: Oxaliplatin — Oxaliplatin 130mg/m2, intravenous drip, on Day 1；
Drug: Capecitabine — Capecitabine 850mg/m2 administrated orally twice daily from Day 1-14.

SUMMARY:
This is an open label, randomized, phase Ⅲ study to treat subjects with RAS/BRAF wild-type, unresectable metastatic colorectal cancer. The patients will be randomized into two arms consist of Anlotinib (3 weeks/cycle) + CapeOx and Bevacizumab (3 week/cycle) + CapeOx at a ratio of 1:1. This study is conducted to assess the efficacy and safety of Anlotinib and Chemotherapy as first-line treatment in subjects with RAS/BRAF wild-type Metastatic Colorectal Cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Understood and Signed an informed consent form. 2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1；Life expectancy≥ 3 months.

  3. Histologically or cytologically confirmed unresectable metastatic colorectal cancer.

  4. Has RAS/BRAF wild-type. 5. Has at least one measurable lesion. 6. Adequate organ function. 7.Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study (such as intrauterine devices , contraceptives or condoms) ; No pregnant or breastfeeding women, and a negative pregnancy test are received within 7 days before the randomization.

Exclusion Criteria:

* 1.Has dMMR/MSI-H. 2. Combined with the following diseases or medical history:

  1. Previous or co-existing malignancies within 3 years except for cured cervical carcinoma in situ, non-melanoma skin cancer and superficial bladder tumors；
  2. Has many factors that affect the oral administration of drugs；
  3. Has Gastrointestinal bleeding or perforation within 4 weeks before the first dose；
  4. Has active inflammatory bowel disease within 4 weeks before the first dose；
  5. Uncontrolled pleural effusion, pericardial effusion or ascites requiring repeated drainage；
  6. Patients whose adverse events (except hair loss) caused by previous treatment did not recover to ≤CTCAE 1 degree；
  7. Has received major surgical procedure、biopsy or obvious traumatic injury within 28 days before the first dose；
  8. Imaging (CT or MRI) shows that tumor invades large blood vessels or the boundary of blood vessels is unclear；
  9. Has any bleeding event or the level of bleeding events ≥ CTCAE 3；
  10. Has unhealed wounds, ulcerative or fractures；
  11. Has arterial or venous thromboembolic events occurred within 6 months, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism；
  12. Has a history of psychotropic substance abuse and are unable to quit ；
  13. Has any severe and / or uncontrolled disease； 3.Tumor related symptoms and treatment

  <!-- -->

  1. Has received chemotherapy, surgery, radiotherapy, and other anti-cancer therapy within 4 weeks before the first dose.
  2. Has received anti-tumor Chinese patent medicine which were approved by NMPA Within 2 weeks before the first dose.
  3. Previous adjuvant therapy containing anti-vascular or anti-EGFR targeted drugs.
  4. Has received systematic treatment for advanced colorectal cancer.
  5. Has symptomatic brain metastases or control of symptoms < 2 month. 4.Has participated in other anticancer drug clinical trials within 4 weeks. 5.According to the judgement of the researchers, there are other factors that may lead to the termination of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 748 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) assessed by IRC | Baseline up to 15 months
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Baseline up to 15 months
  PFS defined as the time from first dose until the first documented progressive disease (PD) or death from any cause.
Overall survival (OS) | Baseline up to 20 months
  OS defined as the time from the first dose to death from any cause. Survival time was censored at the date of last contact for patients who were still alive or lost to follow-up.
Objective Response Rate（ORR） | Baseline up to 15 months
  Percentage of subjects achieving complete response (CR) and partial response (PR) .
Disease Control Rate (DCR) | Baseline up to 15 months
  Percentage of subjects achieving complete response (CR) and partial response (PR) and stable disease (SD).
Duration of Response (DOR) | Baseline up to 15 months
  DOR was defined as the time from the first documentation of objective tumor response (CR or PR) to the first documentation of disease progression or to death due to any cause, whichever occurred first.

CONTACTS AND LOCATIONS:
Locations (92):
- China (92):
  - The People's Hospital of Chizhou, Chizhou, Anhui
  - Fujian Medical University Union Hospital, Fuzhou, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - Anhui Cancer Hospital, Hefei, Anhui
  - Xuancheng People's Hospital, Xuancheng, Anhui
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking University Frist Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fuling Hospital Affiliated to Chongqing University, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - The First Affiliated Hospital Of Guangzhou Medical University, Guangzhou, Guangdong
  - Qingyuan People's Hospital, Qingyuan, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Liuzhou Workers' Hospital, Liuchow, Guangxi
  - The Affiliated Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - The First Hospital of Qinhuangdao, Qinhuangdao, Hebei
  - Tangshan People's Hospital, Tangshan, Hebei
  - The First Affiliated Hospital of Hebei North University, Zhangjiakou, Hebei
  - Harbin Medical University Affiliated Cancer Hospital, Harbin, Heilongjiang
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Huaihe Hospital of Henan University, Kaifeng, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Nanyang Second General Hospital, Nanyang, Henan
  - Xinyang Central Hospital, Xinyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of ZhengZhou University, Zhengzhou, Henan
  - Tongji Hospital Affiliated to Tongji Medical College Hust, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Affiliated Hospital of Chifeng University, Chifeng, Inner Mongolia
  - Chifeng Municipal hospital, Chifeng, Inner Mongolia
  - The First Peoples Hospital of Changzhou, Changzhou, Jiangsu
  - Jiangsu Cancer hospital, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Nanjing Hospital of C.M., Nanjing, Jiangsu
  - Jiangsu Province People's Hospital, Nanjing, Jiangsu
  - Jiangsu Taizhou People's Hospital, Taizhou, Jiangsu
  - Taizhou Second People's Hospital, Taizhou, Jiangsu
  - Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - Subei People's Hospital of Jiangsu Province, Yangzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - JiangXi PingXiang People's Hospital, Pingxiang, Jiangxi
  - Jilin Province FAW General Hospital, Changchun, Jilin
  - Jilin Cancer Hospital, Changchun, Jilin
  - Meihekou Central Hospital, Meihekou, Jilin
  - Yanbian University Hospital, Yanji, Jilin
  - The First Affiliatde Hospital of DaLin Medical University, Dalian, Liaoning
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - Genertec Liaoyou Gem Flower Hospital, Panjin, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Inner Mongolia Autonomous Region Cancer Hospital, Hohhot, Neimenggu
  - Qinghai University Affiliated Hospital, Xining, Qinghai
  - 3201 Hospital, Hanzhong, Shaanxi
  - Hanzhong Central Hospital, Hanzhong, Shaanxi
  - Xi'an International Medical Center Hospital, Xi'an, Shaanxi
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - The Second Affiliated Hospital of PLA Air Force Military Medical University, Xi'an, Shaanxi
  - Shandong Cancer Hospital Affiliated to Shandong Univercity, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Weifang Hospital of Traditional Chinese Medicine, Weifang, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Longhua Hospital Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Changzhi People's Hospital, Changzhi, Shanxi
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Peking University BinHai Hospital, Tianjin, Tianjin Municipality
  - The First People's Hospital of Kashgar, Kashgar, Xinjiang
  - Affiliated Tumor Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Huzhou Cancer Hospital, Huzhou, Zhejiang

REFERENCES:
- [Derived] He J, Liu Y, Liu C, Hu H, Sun L, Xu D, Li J, Wang J, Chen X, Lin R, Jiang Y, Zhang Y, Zhang W, Cheng Y, Wu X, Fang M, Li E, Xu Y, Chen Y, Li J, Cui Y, Pan Z, Zhang S, Yuan Y, Ding K. A Randomized Phase III Study of Anlotinib Versus Bevacizumab in Combination With CAPEOX as First-Line Therapy for RAS/BRAF Wild-Type Metastatic Colorectal Cancer: A Clinical Trial Protocol. Technol Cancer Res Treat. 2023 Jan-Dec;22:15330338231152350. doi: 10.1177/15330338231152350. PMID 36727222